CLINICAL TRIAL: NCT04488172
Title: Exploring the Effects of Genetic Variants and Inflammation on Individualized Treatment Outcomes of Vitamins Supplementation in Patient With Epilepsy
Brief Title: Exploring the Effects of Genetic Variants and Inflammation on Vitamins Supplementation Treatment Outcomes in Epilepsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A-ER-105-489
Record Dates: First submitted 2020-07-21; First posted 2020-07-27 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-02

CONDITIONS: Epilepsy
Keywords: pharmacogenomics; antiepileptic drugs; multi-vitamins supplementation; epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Epilepsy subjects (Experimental): Receiving multi-vitamins supplementation (B6, B9, D, E, Q10) for 6 months trial
  Interventions: Dietary Supplement: Multi-vitamin supplementation

INTERVENTIONS:
Dietary Supplement: Multi-vitamin supplementation — Vitamin B6:100 mg/day Vitamin B9: 5 mg/day Vitamin D: 1000 IU/day Vitamin E: 400 IU/day Co-Q10: 100 mg/day

SUMMARY:
The management of patients with epilepsy is focused on controlling seizures, avoiding treatment side effects, and restoring quality of life. However, about 30% of people are antiepileptic drugs (AEDs) resistance epilepsy after the adequate trials of two AEDs treatment. Genetic factors may contribute to the high interindividual variability in response or adverse effects (such as weight gain and altered lipid profiles) to AEDs. What's more, previous observational studies indicated that vitamin deficiency, such as vitamin B6, is common in patients with epilepsy due to epilepsy itself, AEDs use, or both. Therefore, investigators aim to (1) evaluate the impact of genetic variants on AED and multi-vitamins supplementation in epilepsy, and (2) establish the pharmacogenomics knowledge base of AED and multi-vitamins supplementation on clinical effectiveness in patients with epilepsy.

DETAILED DESCRIPTION:
In the current study, investigators will evaluate the association among the genetic polymorphisms, epilepsy, and multi-vitamins supplementation from Taiwan Biobank and will further investigate potential genes related to vitamins signal pathways (especially vitamin B6, B9, D, E, and Q) involved in epilepsy. These results will not only generate the field of AEDs pharmacogenomics for further study, but also provide new potential treatment targets that may involve in epilepsy therapeutics. The clinical outcomes indicate disease severity, body weight, metabolic indices (i.e., the fasting levels of lipid), HRQoL, anxiety and depression scores. All outcome indicators will be repeated measured at baseline and after 1, 3 and 6 months multi-vitamins supplementation. All of the participants will be assessed the genotypes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic criteria of epilepsy
* Receive anti-epileptic drugs (AEDs)

Exclusion Criteria:

* Have an organic mental disorder, mental retardation, dementia, or other diagnosed neurological illness
* Have a surgical condition or a major physical illness
* Pregnant or breast-feeding

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-04-07 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Seizure severity | 6 months
  Number of seizure attack per month

SECONDARY OUTCOMES:
Medication Compliance | 6 months
  Assessing using Morisky Medication Adherence Scale (MMAS)

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University (NCKU) Hospital, Tainan, Taiwan